CLINICAL TRIAL: NCT03980405
Title: Combination Therapy With Drug and Diet for Induction of Remission in Mild to Moderate Active Pediatric Ulcerative Colitis: A Single Blinded, International Randomized Controlled Trial
Brief Title: Combination of Diet and 5ASA ( 5-aminosalicylic Acid) for Ulcerative Colitis
Acronym: INDUCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It is not possible to continue the study
Sponsor: Prof. Arie Levine (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Arie Levine, Director, Pediatric Gastroenterology and nutrition unit, Wolfson Medical Center
Organization: Wolfson Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001-19-WOMC
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Physicians will be blinded to the randomization and dietary advice received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Control Diet 6 weeks of Oral 5ASA (standard recommended dosing 60-75 mg/kg/day; minimum 2.5, maximum 4 grams/day)+ Low residue diet and 6 more weeks of Oral 5ASA+ Free diet
  Interventions: Dietary Supplement: Group 1- Control Diet
- Group 2 (Experimental): 6 weeks of Oral 5ASA (standard recommended dosing 60-75 mg/kg/day; minimum 2.5, maximum 4 grams/day)+ UC diet and 6 more weeks of Oral 5ASA+ UC diet stage 2
  Interventions: Dietary Supplement: Group 2- UCD Diet

INTERVENTIONS:
Dietary Supplement: Group 1- Control Diet — Oral 5ASA+ Low Residue Diet for 6 weeks and Oral 5ASA+ Free Diet for 6 more weeks
  Arms: Group 1
Dietary Supplement: Group 2- UCD Diet — Oral 5ASA+ UC Diet for 6 weeks and Oral 5ASA+ UC Diet Stage 2 for 6 more weeks
  Arms: Group 2

SUMMARY:
Combination Therapy with Drug and Diet for Induction of Remission in Mild to Moderate Active Pediatric Ulcerative colitis: A Single Blinded, International Randomized Controlled Trial

DETAILED DESCRIPTION:
This will be a 12 week, single blinded Randomized controlled trial (RCT) in children and adolescents with mild to moderate Ulcerative Collitis (UC) comparing 5ASA (recommended dosing 60-75 mg/kg/day; minimum 2.5 maximum 4 grams/day) with fiber restriction for 6 weeks followed by free diet (Group 1) to 5ASA with Ulcerative Collitis Diet (UCD) for 6 weeks, followed by the step down UCD for the next 6 weeks. Inclusion criteria will include children weighing >30kg, Pediatric Ulcerative Collitis Activity index (PUCAI) 10-45, no treatment with 5ASA (treatment naïve or treated with thiopurines for example) or currently treatment with 5ASA but <2 grams/day, ages 10-19 years, with disease extent E2-E4 by the Paris Classification. Patients on thiopurines may continue existing dose if dose is stable for at least 8 weeks.

Exclusion criteria are Patients with acute severe colitis (ASC) in the previous year, requiring oral or intravenous steroids in the previous 3 months, or patients treated with Anti- Tumor necrosis factor alfa (TNFa) regimens. Importantly, there is no placebo arm and both groups will be treated with the same currently recommended drug at currently recommended doses; the only difference between groups being their diets.

The primary endpoint will be remission defined as PUCAI<10 at week 6; Secondary endpoints will be response defined as a drop in PUCAI of 10 or remission at week 6, sustained steroid free remission week 12 and improvement in mucosal healing by Ulcerative Colitis Endoscopic Index of Severity (UCEIS) at week 12 as well as safety and tolerance. Intolerance will be defined as patients stopping the diet because of refusal to continue diet. Patients will be seen at weeks 0, 3, 6, and 12. PUCAI will be assessed at every visit; fecal calprotectin will be assessed at baseline, week 6 and 12. Sigmoidoscopy to assess mucosal healing will be performed at week 12 in patients who had a baseline colonoscopy or sigmoidoscopy. Sigmoidoscopies to evaluate healing will be voluntary and patients will not be excluded if they do not consent to have a follow up sigmoidoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Established diagnosis of UC by the Paris classification and Revised Porto Criteria.
3. Age: 10 - 19 years (inclusive)
4. Mild to moderate active disease, 10 ≤ PUCAI ≤45
5. Extent E2-E4 by the Paris classification
6. Weight >30 kg (ensures that patients who received 5ASA ≤2 grams are eligible)
7. Stable medication (IMM/ 5ASA) use or no change in medication use for the past 6 weeks. Patients who have received topical 5ASA therapy for <10 days and are active may be included if topical therapy is stopped at enrolment.
8. Patients not receiving 5ASA or using 5ASA<50mg/kg/day

Exclusion Criteria:

1. Any proven current infection such as positive stool culture, parasite or C. difficile.
2. Steroids (oral or intravenous) use in the past 3 months.
3. Patients who continue topical 5ASA or steroids after enrolment
4. Use of biologics in present or in past 6 months
5. Use of antibiotics for more than one week in the past 60 days
6. PUCAI >45
7. Acute severe UC in the previous 12 months.
8. Current extra intestinal manifestation of UC.
9. Primary Sclerosing Cholangitis (PSC) or Liver disease
10. Pregnancy.
11. Vegans or patients unwilling or unable to consume eggs
12. Inflammatory Bowel Disease (IBD) unclassified

Exclusion criteria Comments:

1. Stool culture, parasite or C. difficile will only be measured if the patient has diarrhea.
2. Patients who have received treatment enemas for 3 weeks or less then 3 days and are active, can be included but must stop the enemas on the day of enrolment

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
PUCAI< 10 at week 6 | 6 weeks
  Remission defined as PUCAI<10 at week 6

SECONDARY OUTCOMES:
A drop of PUCAI at least 10 points or remission | 6 weeks
  Response defined as a drop of PUCAI at least 10 points or remission (intention to treat) week 6 .
Mean/median change in Calprotectin at week 6 | 6 weeks
  Mean/median change in Calprotectin at week 6
Sustained remission week 12 | 12 weeks
  Sustained steroid & biologic free remission week 12
Need for topical therapy by week 12 | 12 weeks
  Need for topical therapy by week 12
Change in UCEIS at week 12 ( optional) | 12 weeks
  Change in UCEIS at week 12 ( optional)
Tolerance to diet | 12 weeks
  Tolerance to diet defined by withdrawal from the study because of difficulties with the diet.

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, Prof, Principal Investigator — Wolfson Medical Center
Locations (1):
- Wolfson MC, Holon, Israel

IPD SHARING:
Plan to Share IPD: No